CLINICAL TRIAL: NCT02022774
Title: A Single-arm, Open, Clinical Study to Evaluate the Effects of Fimasartan on Arterial Stiffness in Patients With Hypertension
Brief Title: Efficacy of fimaSartan on arTerIal stiFFness iN patiEntS With HypertenSion
Acronym: STIFFNESS
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CN-KKH-01
Record Dates: First submitted 2013-12-03; First posted 2013-12-30 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — fimasartan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fimasartan — Fimasartan 60 ~ 120 mg/po take one tablet once a day
  Other Names: BR-A-657-K

SUMMARY:
The purpose of this study is to evaluate the effects of fimasartan on arterial stiffness in patients with hypertension

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to participate in this study and give written informed consent
* Subjects whose sitting diastolic blood pressure measured at placebo visit and baseline are more than 90 mmHg and/or systolic blood pressure are more than 140 mmHg
* Subjects who are naive to anti-hypertensive treatment
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

* Subjects who are hypersensitive to angiotensin type 1-receptor blockers
* Subjects with secondary hypertension
* Subjects with severe hypertension (systolic blood pressure >= 180 mmHg OR diastolic blood pressure >= 110)
* Severe cardiac disease (heart failure, ischemic heart disease, peripheral vascular disease, moderate valvular disease, arrhythmia requiring treatment, cardiomyopathy, etc.)
* Subjects with chronic obstructive pulmonary disease or history
* Clinically significant renal dysfunction (Creatinine 2.0 mg/dL) and liver dysfunction (ALT, AST > 2x UNL)
* Subjects with life expectancy of less than 2 years due to non-cardiac disease
* Subjects with history or evidence of abuse of drugs or alcohol within 2 years
* Severe insulin-dependent diabetes mellitus or intractable diabetic patient (dose/regimen change of oral hypoglycemic agent, insulin use)
* Severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, within 6 months)
* Wasting diseases, autoimmune diseases (rheumatoid arthritis, systemic lupus anticoagulants, etc.), history of connective tissue disease or ongoing disease.
* Women with pregnancy and breast feeding
* Women planning to be pregnant or without admitted contraception despite of probability of pregnancy (Women who underwent sterilization operation are excluded. Fertile women without such surgery should undergo pregnancy test and can participate only with negative result. Intermittent abstinence like basic body temperature method, natural period method are not considered admitted contraception and no hormonal contraception is allowed.).
* Subjects who are participating in other clinical trials for investigating agents or have taken other clinical trial medication within 4 weeks before screening visit.
* Subjects judged to be inappropriate by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple secondary and tertiary centers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement of carotid radial strain value | 24 weeks
  Improvement of carotid arterial stiffness measured by echocardiography

SECONDARY OUTCOMES:
Improvement in brachial-ankle pulse wave velocity (baPWV) | 24 weeks
Improvement in augmentation index (AIx) | 24 weeks
Improvement in carotid distensibility | 24 weeks
Improvement in sitting systolic blood pressure (SiSBP) | 24 weeks
Improvement in sitting diastolic blood pressure (SiDBP) | 24 weeks
Improvement in central blood pressure (BP) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kye Hun Kim, MD, Principal Investigator — Chonnam National University Hospital
Locations (7):
- South Korea (7):
  - St. Carollo Hospital, Suncheon, Jeollanamdo
  - Chonnam National University Hospital, Gwangju
  - Gwagnju Christian Hospital, Gwangju
  - Gwanju Veterans Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Jeonbuk National University Hospital, Jeonju
  - Jeonju Jesus Hospital, Jeonju